CLINICAL TRIAL: NCT02991716
Title: Surface Electrocardiogram (ECG) Signal Recording for Implantable Subcutaneous String Defibrillator (ISSD) Development
Status: Completed | Type: Observational
Sponsor: NewPace Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NPC02
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Arrhythmia, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recorded patients: Patients requiring Intracradiac Defibrillator (ICD) implantation, Electrophysiology (EP) study or a holter monitor recording, mainly due to suspected ventricular tachy - arrhythmias
  Interventions: Other: recorded patients

INTERVENTIONS:
Other: recorded patients — No intervention applied, only recording of cutaneous ECG signal from specific points on the torsi

SUMMARY:
Record cutaneous Electrocardiogram (ECG) data from positions corresponding to the expected subcutaneous locations of the Implantable Subcutaneous String Defibrillator (ISSD) using existing, approved ECG recording devices.

DETAILED DESCRIPTION:
2 electrodes places near the sternum and 2 near the midaxillary line, simulating the expected positions of Implantable Subcutaneous String Defibrillator (ISSD) sense electrodes. reference ECG electrodes are also attached (in most cases). Approved ECG recording devices are used to record the signal continuously: During an EP session (different types) a bedside recorder, and a holter monitor is used during holter recordings. Ep session recordings are performed in order to capture different types of arrhythmia, and holter recordings are performed to observe changes in ECG morphology due to activity, position changes, circadian cycles etc. The data is saved and used in the development of the ISSD.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ICD implantation
* Candidate for EP study
* Candidate for 24 hour holter monitor recording

Exclusion Criteria:

* age<18

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring Intracradiac Defibrillator (ICD) implantation, Electrophysiology (EP) study or a holter monitor recording, mainly due to suspected ventricular tachy - arrhythmias
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
successful recording of Electrocardiogram (ECG) from a patient containing arrhythmia | immediate
  recorded Electrocardiogram (ECG) of patients with as many arrhythmia events as possible, preferably tachy-arrhythmia events such as fast VT, flutter or VF

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Rankovic, M.D, Principal Investigator — JFK Medical Center, Florida
Locations (1):
- JFK Medical Center, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No